CLINICAL TRIAL: NCT06302764
Title: Analysis of the Occupational Workload of Doctors and Medical Staff Involved in Emergency and Life-threatening Situations
Brief Title: Emergency Medical Staff Workload Analysis
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Krystyna Golonka, Professor, Jagiellonian University
Other Study IDs: WZiKS.4.1.2023.2; WZiKS.4.1.2023 (Other Grant/Funding Number: Jagiellonian University in Kraków)
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Stress; Work Related Stress; PTSD; Mental Stress; Medical Emergencies
Keywords: stress; work-related stress; trauma; PTSD; medical personnel
MeSH Terms: conditions — Occupational Stress; Stress Disorders, Post-Traumatic; Stress, Psychological; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Polish Medical Staff: Medical doctors, and emergency staff (paramedics), involved in treating life-threatening conditions
  Interventions: Diagnostic Test: Qualitative & Quantitative Research
- Ukrainian Medical Staff: Medical doctors, and emergency staff (paramedics), involved in treating life-threatening conditions
  Interventions: Diagnostic Test: Qualitative & Quantitative Research
- Portuguese Medical Staff: Medical doctors, and emergency staff (paramedics), involved in treating life-threatening conditions
  Interventions: Diagnostic Test: Qualitative & Quantitative Research
- Spanish Medical Staff: Medical doctors, and emergency staff (paramedics), involved in treating life-threatening conditions
  Interventions: Diagnostic Test: Qualitative & Quantitative Research

INTERVENTIONS:
Diagnostic Test: Qualitative & Quantitative Research — 1. Focused interviews - conducted by members of the appointed research team to recognize the issues faced by emergency medical staff in Poland, Ukraine, Portugal, and Spain with the aim of preparing the measurement framework.
  2. Online questionnaire surveys - conducted using the Qualtrics platform (available in different, language versions - Polish, Ukrainian, Portuguese, and Spanish).

SUMMARY:
The aim of this study is to identify trauma determinants and leverage this understanding to develop solutions applicable to the prevention and treatment of PTSD among emergency medical personnel. By categorizing stimuli associated with traumatic professional experiences, the study aims to enhance existing therapeutic protocols through exposure therapy. The specific objectives are as follows:

1. Analysis and characterization of occupational workloads among doctors and emergency medical personnel, focusing on the scale of burdens associated with PTSD symptoms.
2. Development of categories for aggravating and potentially traumatizing stimuli within the medical staff of rescue teams.
3. Examination of the feasibility of incorporating the obtained results into cognitive-behavioral therapy protocols.
4. Assessment of the potential for implementing the results in solutions utilizing virtual reality technology.
5. Formation of an interdisciplinary international research team.

DETAILED DESCRIPTION:
Background: Data on the impact of workloads indicate that emergency medical personnel exposed to sudden threats to health or life are particularly vulnerable to the consequences of occupational stress. Symptoms of Post-Traumatic Stress Disorder (PTSD) within this professional group significantly surpass the rates found in the general population. Traumatic experiences encountered by medical staff may lead to a substantial decline in their mental health, as well as in their social and professional functioning.

Participants: Several hundred medical doctors and emergency medical personnel from Poland, Ukraine, Portugal and Spain.

Research Methodology: Analysis of data collected through focused interviews, psychological scales, and questionnaires pertaining to burnout, stress, and mental health conditions.

ELIGIBILITY:
Inclusion Criteria:

* completed medical studies or emergency medical course
* assistance in life-threatening conditions

Exclusion Criteria:

* Intellectual disability
* Inability to self-complete the research questionnaires

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff involved in treating life-threatening conditions
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Focused Interview | October, 2023 until November, 2023
  Interviews pertaining to physical injury risk, psychosocial factors, and personal indicators
Posttraumatic Stress Disorder Checklist (PCL-5) | December, 2023 until March, 2024
  Posttraumatic Stress Disorder Checklist - 20-item, self-report measure to assess the symptoms of posttraumatic stress disorder. Items are rated on 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely). A general score ranges from 0 to 80 with a higher score indicating a higher symptoms of posttraumatic stress disorder.
Patient Health Questionnaire (PHQ-9) | December, 2023 until March, 2024
  Patient Health Questionnaire - 9-item, self-report measure to assess the severity of depression. Items are rated on 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). A general score ranges from 0 to 27 with a higher score indicating a higher depressive symptom severity.
Depersonalization Mechanism Scale (DMS) | December, 2023 until March, 2024
  Depersonalization Mechanism Scale - a 20-item, self-report measure to assess the tendency to depersonalization. Items are rated on 5-point Likert scale, ranging from 0 (never) to 4 (very often). A general score ranges from 0 to 80 with a higher score indicating a higher tendency to depersonalization.

CONTACTS AND LOCATIONS:
Overall Officials: Krystyna Golonka, Prof, Principal Investigator — Jagiellonian University
Locations (3):
- Institute of Applied Psychology, Jagiellonian University in Krakow, Poland, Krakow, Małopolska, Poland
- University of Coimbra, Coimbra, Portugal
- Bogomolets National Medical University, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided